CLINICAL TRIAL: NCT03018184
Title: Contractile Cross Sectional Areas and Muscle Strength in Patients With Congenital Myopathies Compared to Healthy Controls
Brief Title: Contractile Cross Sectional Areas and Muscle Strength in Patients With Congenital Myopathies
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Anne-Sofie Vibæk Eisum, BSc Med., Rigshospitalet, Denmark
Other Study IDs: H-16045346
Record Dates: First submitted 2017-01-10; First posted 2017-01-11 (Estimated); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Inherited Muscle Diseases; Congenital Myopathy; RYR1-myopathy
Keywords: MRI; CCSA; Contractile Cross Sectional Area; Strength
MeSH Terms: conditions — Myotonia Congenita | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: MRI and Muscle Dynamometer

SUMMARY:
Patients with inherited muscle diseases can have several problems in their muscles, which can be both structural and metabolic. All the different diseases can affect the contractility of the muscles. The aim of the study is to investigate the relation between muscle strength and contractile cross sectional area (CCSA) in the thigh and calf in patients affected by inherited muscle diseases.

DETAILED DESCRIPTION:
Patients with inherited muscle diseases can have several miscellaneous problems in their muscles, which can be both structural and metabolic. Depending on the specific disease multiple symptoms may be present. All the different diseases can affect the contractility of the muscles. Examples of inherited muscle diseases are congenital myopathies and RYR1-myopathy, afflicting the muscle fiber structure. They are the first subgroups of inherited muscle diseases to be investigated in this study. Congenital myopathies are hereditary and relatively non-progressive diseases. Hypotonia is the clinical characteristic of congenital myopathies and is often presented already in the neonatal period. Almost all patients have generalized muscle weakness and hypotonia. The various subtypes of congenital myopathy are a broad group of disorders defined by the predominance of particular and specific structural abnormalities shown in muscle biopsies. Based on genetic and morphological features, they can be divided into four main groups; one with central cores, one with central nuclei, one with minicores and one with nemaline bodies. RYR1-myopathy is caused by a mutation in the RYR-gene. The RYR1-protein is important in the making of RYR1-receptors and channels responsible for the transport of calcium atoms within muscle cells, particularly in muscle contractions. Patients typically present with limb weakness, decreased fetal movement and skeletal abnormalities. About 70% of patients with malignant hyperthermia have a mutation in the RYR1-gene. MRI findings often include involvement of different muscles in the thigh and the calf.

ELIGIBILITY:
Inclusion Criteria:

* Verified inherited muscle disease.
* Age: Over 18 years old

Exclusion Criteria:

* Contraindications for an MRI.
* Claustrophobia.
* Pregnant or nursing women.
* Competing disorders (as arthritis) or other muscle disorders.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with verified inherited muscle disease.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2016-12; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Muscle CCSA, investigated by Dixon MRI techniques. | MRI scan per subject lasts approximately 60 minutes.
  The MRI protocol include a whole body scan. The calf and thigh are chosen for qualitative analysis. Cross sectional area is calculated, the amount of adipose tissue is calculated, and the amount of adipose tissue is subtracted from the CSA, resulting in the CCSA.
Muscle strength, measured as peak torque, investigated by an isokinetic dynamometer (Biodex 4). | The tests takes less than an hour per subject.
  The dynamometer makes it possible to isolate particular muscle groups. It is possible to control the range of motion and thereby test in an area free of pain.

SECONDARY OUTCOMES:
Muscle Strength, MRC | The exam lasts less than 15 min per subject.
  Assessment of the muscle strength by a clinical test using "the Medical Research Council Scale for muscle strength" (MRC-scale).

CONTACTS AND LOCATIONS:
Overall Officials: John Vissing, MD DMSc, Principal Investigator — Copenhagen Neuromuscular Center, Rigshospitalet
Locations (1):
- Copenhagen Neuromuscular Center, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Congenital Myopathies: Background, Pathophysiology, Epidemiology [Internet]. [henvist 18. oktober 2016]. Tilgængelig hos: http://emedicine.medscape.com/article/1175852-overview
- [Background] Hilton-Jones D, Martin R. Turner. Oxford Textbook of Neuromuscular Disorders. I: Oxford Textbook of Neuromuscular Disorders. Oxford; s. 277-87.
- [Background] Congenital Myopathies Clinical Presentation: History, Causes [Internet]. [henvist 18. oktober 2016]. Tilgængelig hos: http://emedicine.medscape.com/article/1175852-clinical
- [Background] Paternostro-Sluga T, Grim-Stieger M, Posch M, Schuhfried O, Vacariu G, Mittermaier C, Bittner C, Fialka-Moser V. Reliability and validity of the Medical Research Council (MRC) scale and a modified scale for testing muscle strength in patients with radial palsy. J Rehabil Med. 2008 Aug;40(8):665-71. doi: 10.2340/16501977-0235. PMID 19020701
- [Background] Lokken N, Hedermann G, Thomsen C, Vissing J. Contractile properties are disrupted in Becker muscular dystrophy, but not in limb girdle type 2I. Ann Neurol. 2016 Sep;80(3):466-71. doi: 10.1002/ana.24743. Epub 2016 Aug 10. PMID 27463532